CLINICAL TRIAL: NCT06944899
Title: A Single-Center Pilot Study to Test the Effectiveness of the REPAIR Nitric Oxide (NO) Sensor to Record Wound Characteristic Data
Brief Title: NO Sensor to Record Wound Data in Acute or Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Badylak (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Stephen Badylak, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY25010133; D20AC00002-13 (Other Grant/Funding Number: DARPA)
Record Dates: First submitted 2025-04-04; First posted 2025-04-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Volumetric Muscle Loss

STUDY DESIGN:
Intervention Model Description: proof of concept
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NO Sensor (Experimental): NO sensor placed into wound bed
  Interventions: Device: NO Sensor

INTERVENTIONS:
Device: NO Sensor — NO sensor measuring wound characteristic data in wound bed

SUMMARY:
The purpose of this research is to evaluate the ability of a Nitric Oxide (NO) Sensor to collect NO measurement data from an open wound. Previous research suggests that NO levels may indicate the stage of healing the wound is in. This study is being done to determine if the NO Sensor can measure how much NO is in a participant's wound. The researcher will place the NO Sensor into a participant's wound to collect NO measurements for 30-60 minutes. The participant will then have 2 follow-up appointments to see how the wound heals over time.

ELIGIBILITY:
Inclusion Criteria:

1. Extremity injury
2. Wound surface area 2-10 cm in diameter
3. Wound amenable to NO Sensor placement
4. Age at the time of consent ≥ 22 to ≤ 65 years
5. Cognitively able to undergo informed consent discussion and understand the study

Exclusion Criteria:

1. Chemotherapy
2. Pregnancy
3. Preexisting immunosuppressive conditions or immunosuppression therapy
4. Active hemorrhage in the wound bed
5. Physician discretion for patients with complex medical conditions or high mortality risks
6. Patients with an active implanted device, such as a pacemaker, defibrillator, or hypoglossal or vagal nerve stimulator
7. Patients requiring a legally authorized representative (LAR) for informed consent

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Participants meet all inclusion/exclusion criteria - a minimum of 5 participants have completed Inclusion/Exclusion in CRF-01 | up to 8 weeks
All wound characteristics documented - a minimum of 5 wounds assessed by Bates-Jensen Wound Assessment Tool. And documented in CRF-03 | Day 0
NO Sensor application time > 30 minutes and < 60 minutes - a minimum of 5 wounds have NO sensor applied between 30-60 minutes and documented in CRF-04 | 60 minutes
NO Sensor applied and removed according to study specific SOPs - a minimum of 5 wounds have NO Sensor applied and removed according to study specific SOPs and documented in CRF-04 | Day 0
Assessment of wound healing during participant follow-up activities - a minimum of 5 participants have follow up wound assessments according to visit schedule and documented in CRF-05 and CRF-06 | up to 8 weeks
  A follow up phone call within 72 hours and an in-person clinic visit within 2-8 weeks of NO Sensor application

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Badylak, MD,DVM,PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Mercy, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
no plan to raw share data